CLINICAL TRIAL: NCT00389610
Title: A Safety and Efficacy Trial of Vaccine Boosting With Lethally Irradiated Allogeneic Pancreatic Tumor Cells Transfected With the GM-CSF Gene for the Treatment of Pancreatic Adenocarcinoma
Brief Title: Adjuvant GVAX Vaccine Therapy in Patients With Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: The Skip Viragh Foundation (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J0619; P30CA006973 (NIH); JHOC-SKCCC-J0619 (JHM IRB); NA_00002731
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Results first posted 2022-09-02 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Pancreatic Cancer
Keywords: stage I pancreatic cancer; stage II pancreatic cancer; pancreatic neoplasm; adenocarcinoma of the pancreas; stage IIl pancreatic cancer; adjuvant therapy; cancer vaccine; GVAX
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Previously Vaccinated With GVAX Pancreas Vaccine (Experimental): Participants receive booster vaccination every 6 months, given intradermally.
  Interventions: Biological: GVAX pancreas vaccine
- GVAX Pancreas Vaccine Naive (Experimental): Participants will receive GVAX pancreas priming vaccinations once every month for a total of 3 months and every 6 months after that, given intradermally.
  Interventions: Biological: GVAX pancreas vaccine

INTERVENTIONS:
Biological: GVAX pancreas vaccine — Given intradermally
  Other Names: Two irradiated allogeneic pancreatic tumor cells transfected with the GM-CSF gene

SUMMARY:
This is an open label, phase II trial study of adjuvant GVAX pancreas vaccine in patients with pancreatic cancer.

DETAILED DESCRIPTION:
Eligible participants will receive by intradermal administration the GVAX pancreas vaccine consisting of two irradiated allogeneic pancreatic tumor cell lines transfected with the granulocyte macrophage-colony stimulating factor (GM-CSF) gene.

There will be two cohorts of research participants:

1. Participants previously vaccinated with GVAX pancreas vaccine. These participants will receive booster vaccinations as a continuation of care. Vaccination repeats every 6 months in the absence of disease progression or unacceptable toxicity.
2. Participants who were not previously vaccinated with GVAX pancreas vaccine (vaccine naive). These participants received priming vaccinations once a month for 3 months followed by booster vaccinations every 6 months.

ELIGIBILITY:
1. Inclusion Criteria:

   A. previously vaccinated subjects must receive Gvax vaccine previously

   B. naïve and previously vaccinated subjects must meet the following criteria:
   * have a history of surgically resected pathologic stage 1,2 or 3 adenocarcinoma of the head, neck, tail, or uncinate of the pancreas
   * received the last anti-cancer therapy at least 28 days ago.
   * provide informed consent.
   * have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
   * have adequate hematologic function (Hemoglobin ≥ 9 gm/dl, Absolute neutrophil count (ANC) ≥ 1500 #/cu mm, platelets ≥100,000 K/cu mm)
   * have adequate renal function (Serum creatinine ≤ 2 mg/dL).
   * have adequate hepatic function (Bilirubin ≤ 2.0 mg/dL, unless known Gilbert's Syndrome; Aspartate Aminotransferase (AST), Alanine transaminase (ALT) and amylase ≤ 2x upper limit of normal: Alk Phosphatase ≤ 5x upper limit of normal.)
   * agree to use adequate birth control, if of childbearing potential.
2. Exclusion criteria:

   * radiographical evidence of pancreatic cancer disease recurrence
   * documented history of autoimmune diseases including systemic lupus erythematosus, sarcoidosis, rheumatoid arthritis, glomerulonephritis, or vasculitis
   * uncontrolled medical problems
   * systemic steroid therapy within 28 days before vaccine administration
   * anticipated need for systemic steroid therapy within 28 days after vaccine administration
   * evidence of active infections
   * pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2006-09-11 (Actual); Primary Completion 2021-10-11 (Actual); Study Completion 2022-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A. Laheru, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Previously Vaccinated With GVAX Pancreas Vaccine | GVAX Pancreas Vaccine Naive
Started | 11 | 45
Completed | 11 | 23 (milestone period is defined as receiving at least one booster vaccine)
Not Completed | 0 | 22
Not completed — Disease Progression | 0 | 19
Not completed — Death | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Previously Vaccinated With GVAX Pancreas Vaccine | GVAX Pancreas Vaccine Naive | Total
Number analyzed (Participants) | 11 | 45 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 29 | 30
  >=65 years | 10 | 16 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 19 | 23
  Male | 7 | 26 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 10 | 44 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 9 | 42 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Experiencing a Grade 3 or Above Treatment- Related Toxicity
Description: When calculating the incidences of adverse events, each adverse event (as defined by NCI CTCAE v3) will be counted only once for a given subject.
Time Frame: 14 years
Measure: Count of Participants; unit: Participants
Arm/Group | Previously Vaccinated With GVAX Pancreas Vaccine | GVAX Pancreas Vaccine Naive
Number analyzed (Participants) | 11 | 45
Participants | 1 | 5

2. Secondary Outcome: Overall Survival (OS)
Description: OS will be measured from date of first dose until death or end of follow-up (OS will be censored on the date the subject was last known to be alive for subjects without documentation of death at the time of analysis). Estimation based on the Kaplan-Meier curve.
Time Frame: 16 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Previously Vaccinated With GVAX Pancreas Vaccine | GVAX Pancreas Vaccine Naive
Number analyzed (Participants) | 11 | 45
Months | 80.5 [22.5 to 187.8] | 30.7 [19.3 to 40.7]

3. Secondary Outcome: Disease-free Survival (DFS)
Description: DFS is defined as the time from the first dose until evidence of disease recurrence or progression confirmed by first scan. DFS will be censored at the date of the last scan for subjects without documentation of disease recurrence or progression at the time of analysis. Estimation based on the Kaplan-Meier curve.
Time Frame: 16 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Previously Vaccinated With GVAX Pancreas Vaccine | GVAX Pancreas Vaccine Naive
Number analyzed (Participants) | 11 | 45
Months | 109.5 [5.59 to NA] — NA Explanation: Upper bound confidence interval was not reached. | 13.7 [5.55 to 25.1]

ADVERSE EVENTS:
Time Frame: 16 years
Description: This study used the descriptions and grading scales found in the revised National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 for adverse event reporting. During the survival follow-up portion of the trial, patients were evaluated for all-cause mortality past the time frame for treatment and the assessment of adverse events. Adverse events were assessed for up to 14 years. All-Cause Mortality was assessed for up to 16 years.
Arm/Group | Previously Vaccinated With GVAX Pancreas Vaccine | GVAX Pancreas Vaccine Naive
All-Cause Mortality (participants affected / at risk) | 10/11 | 42/45
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/45
Other Adverse Events (participants affected / at risk) | 11/11 | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Previously Vaccinated With GVAX Pancreas Vaccine (N=11) | GVAX Pancreas Vaccine Naive (N=45)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Previously Vaccinated With GVAX Pancreas Vaccine (N=11) | GVAX Pancreas Vaccine Naive (N=45)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 3 (4)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Chills (General disorders) | 4 (7) | 6 (6)
Fatigue (General disorders) | 2 (3) | 10 (14)
Fever (General disorders) | 1 (1) | 6 (16)
Flu-Like symptoms (General disorders) | 9 (23) | 23 (62)
Malaise (General disorders) | 0 (0) | 4 (4)
White blood cell count elevated (Investigations) | 1 (1) | 3 (4)
Eosinophil count elevated (Investigations) | 1 (1) | 16 (16)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 8 (8)
Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 4 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Blisters (Skin and subcutaneous tissue disorders) | 3 (8) | 8 (13)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (5)
Urticaria (Skin and subcutaneous tissue disorders) | 4 (10) | 10 (17)
Bruising (vaccination site) (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Erythema (vaccination site) (Skin and subcutaneous tissue disorders) | 11 (64) | 45 (250)
Vaccine Flares (vaccination site) (Skin and subcutaneous tissue disorders) | 4 (18) | 13 (38)
Induration (vaccination site) (Skin and subcutaneous tissue disorders) | 11 (64) | 45 (247)
Skin hyperpigmentation (vaccination site) (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (7)
Tenderness (vaccination site) (Skin and subcutaneous tissue disorders) | 9 (56) | 34 (146)
Pruritus (vaccination site) (Skin and subcutaneous tissue disorders) | 11 (53) | 37 (191)
Warmth (vaccination site) (Skin and subcutaneous tissue disorders) | 10 (42) | 35 (87)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-07): https://cdn.clinicaltrials.gov/large-docs/10/NCT00389610/Prot_SAP_000.pdf